CLINICAL TRIAL: NCT02447419
Title: Study to Evaluate the Safety and Efficacy of Gefitinib, in Subjects With EFGR Amplification Refractory Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, MD,PhD, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-10-029
Record Dates: First submitted 2015-05-14; First posted 2015-05-18 (Estimated); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gefitinib (Experimental): Gefitinib 250 mg will be administered orally daily
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: Gefitinib — Gefitinib 250mg will be administered orally daily

SUMMARY:
This study is a single-arm,phase II study of gefitinib in patient with epidermal growth factor receptor amplification Refractory solid tumors.

Gefitinib 250 mg will be administered orally daily.

To investigate the efficacy and safety of gefitinib in patient with epidermal growth factor receptor amplification Refractory solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of fully informed consent prior to any study specific procedures.
2. Patients must be ≥20 years of age.
3. Patient with Epidermal growth factor receptor amplification Refractory Solid Tumors and/or specific sensitivity to Gefitinib by Avatar scan that has recurred or progressed following standard therapy, or that has not responded to standard therapy, or for which there is no standard therapy.

   (EGFR amplification by cancer scan + EGFR IHC overexpression +2 or +3)
4. ECOG performance status 0-2.
5. Have measurable or evaluated disease based on RECIST1.1. as determined by investigator.
6. Adequate Organ Function Laboratory Values

   * Absolute neutrophil count ≥ 1.5 x 109/L, Hemoglobin ≥ 9g/dL, Platelets ≥ 100 x 109/L
   * bilirubin ≤ 1.5 x upper limit of normal AST/ALT ≤ 2.5 x upper limit of normal (5.0 X upper limit of normal , for subjects with liver metastases)
   * creatinine ≤1.5 x UNL
7. Patients of child-bearing potential should be using adequate contraceptive measures (two forms of highly reliable methods) should not be breast feeding and must have a negative pregnancy test prior to start of dosing.
8. Adequate heart function.

Exclusion Criteria:

1. Patients with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≤5 years.
2. Has known active central nervous system (CNS) metastases.
3. Has an active infection requiring systemic therapy.
4. Pregnancy or breast feeding
5. Patients with cardiac problem.
6. KRAS mutation (codon 12 or 13) or BRAF mutation (V600)
7. Any previous treatment with Gefitinib
8. Patients with a risk factor of interstitial lung disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-12-03 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
overall response rate | up too 100 weeks

SECONDARY OUTCOMES:
progression-free survival | expected average of 24 weeks
overall survival | up too 100 weeks
Number of subjects with Adverse Events as a measure of safety | up too 100 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Byeon S, Hong JY, Lee J, Nam DH, Park SH, Park JO, Park YS, Lim HY, Kang WK, Kim ST. Use of Gefitinib in EGFR-Amplified Refractory Solid Tumors: An Open-Label, Single-Arm, Single-Center Prospective Pilot Study. Target Oncol. 2020 Apr;15(2):185-192. doi: 10.1007/s11523-020-00706-0. PMID 32107712